CLINICAL TRIAL: NCT03956186
Title: Can we Predict Predict Spinal Anesthesia Induced Hypotension During Caesarean Section Using Right Toe Perfusion Index or Pleth Variability Index?
Brief Title: Can Right Toe Perfusion Index or Pleth Variability Index Predict Spinal Anesthesia Induced Hypotension?
Status: Completed | Type: Observational
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Responsible Party: Principal Investigator, MAHMUT ARSLAN, Assistant Professor, Kahramanmaras Sutcu Imam University
Other Study IDs: KSU 2019-07
Record Dates: First submitted 2019-05-16; First posted 2019-05-20 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Cesarean Section Complications; Hypotension; Spinal Anesthesia; Perfusion Index; Pleth Variability Index
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypotension group: Parturients undergoing elective C/S under spinal anesthesia whose systolic arterial pressure drop below 80 mmHg or have symptoms of hypotension such as dizziness, nausea and vomiting during the procedure.
- Non-hypotension group: Parturients undergoing elective C/S under spinal anesthesia whose systolic arterial pressure does not drop below 80 mmHg or have any symptoms of hypotension during the procedure.

SUMMARY:
Spinal anesthesia for caesarean section is associated with a decrease in systemic vascular resistance and cardiac output and may cause hypotension in a significant portion of the parturients. Hypotension during delivery may cause maternal and fetal complications. If parturients who are likely to develop hypotension after spinal anesthesia can be identified before surgery, anesthesiologists would have opportunity to take measures such as prophylactic vasopressor administration. Perfusion index (PI) measured by pulse oximetry reflects vasomotor tone which affects the degree of hypotension after spinal anesthesia. This is a non-invasive method of assessing the relative vascular tone with the use of pulse oximeter which calculates the ratio of pulsatile versus the non-pulsatile component of the blood flow. A lower PI indicates greater peripheral vasomotor tone. Pleth variability index (PVI) is calculated using maximum and minimum values of perfusion index during respiratory cycles. PVI is one of the dynamic indices that can predict fluid responsiveness. There are several studies investigating the predictive value of finger PI and PVI on hypotension after spinal anesthesia. However the aortocaval compression by the gravid uterus directly effects the lower extremity perfusion. So, in this study we aimed to investigate whether the right toe PI and PVI values at supine and left lateral positions can predict hypotension during caesarean section.

ELIGIBILITY:
Inclusion Criteria:

* singleton parturient
* planned for elective LSCS under spinal anesthesia

Exclusion Criteria:

* gestational age < 36 weeks

  * emergency cases
  * placenta previa, pre-eclampsia
  * BMI>40
  * Reynauld disease
  * patient refusal
  * cardiovascular disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Parturients scheduled for elective low segment caesarean section under spinal anesthesia
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
pleth variability index (PVI) | perioperative
  PVI values (%)at supine and lateral positions, before and after spinal anesthesia will be recorded and compared between the 2 groups.
Perfusion index (PI) | perioperative
  PI values(%)at supine and lateral positions, before and after spinal anesthesia will be recorded and compared between the 2 groups.

SECONDARY OUTCOMES:
blood pressure (mmHg) | perioperative
  blood pressure will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: MAHMUT ARSLAN, Study Director — KSU school of medicine
Locations (1):
- Kahramanmaras Sutcu Imam University, Kahramanmaraş, In the USA Or Canada, Please Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No